CLINICAL TRIAL: NCT00796393
Title: Effects of Daily Consumption of a Probiotic on the Evolution of Infectious Episodes (ENT, Gastro-intestinal and Pulmonary), in Subject Aged 60 Years or Over, During Winter.
Brief Title: Study of the Effects of Probiotics Upon Infectious Episodes in Subject Aged More Than 60, During Winter.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Rosell Lallemand (Industry)
Collaborators: BioFortis (Other)
Responsible Party: Henri Durand, Institut Rosell Lallemand
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 10308; 2008-A01187-48
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Infectious Episodes (ENT, Gastro-intestinal and Pulmonary)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2 (Experimental): Subject with active product, not vaccinated against influenza.
  Interventions: Dietary Supplement: Lactobacillus helveticus R0052, Bifidobacterium bifidum R0071, Bifidobacterium infantis R0033
- 3 (Placebo Comparator): Subject with placebo, vaccinated against influenza.
  Interventions: Dietary Supplement: Starch of potato
- 4 (Placebo Comparator): Subject with placebo, not vaccinated against influenza.
  Interventions: Dietary Supplement: Starch of potato
- 1 (Experimental): Subject with active product, vaccinated against influenza
  Interventions: Dietary Supplement: Lactobacillus helveticus R0052, Bifidobacterium bifidum R0071, Bifidobacterium infantis R0033

INTERVENTIONS:
Dietary Supplement: Lactobacillus helveticus R0052, Bifidobacterium bifidum R0071, Bifidobacterium infantis R0033 — 1 pill per day for 12 weeks
  Arms: 1; 2
Dietary Supplement: Starch of potato — 1 pill per day for 12 weeks
  Arms: 3; 4

SUMMARY:
We put forward that probiotics have an effect on infectious episodes evolution in subjects aged 60 years or over. The main objective of this research is to observe the effect of consumption of the probiotic on the average number of days with infectious episodes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who accept not to alter their food habits

Exclusion Criteria:

* Food allergy
* Regular consumption of probiotics
* Diabetes
* Respiratory deficiency
* Cardiac deficiency
* Cancer or chronicle disease not stabilized
* Splenectomy, sickle-cell anemia
* Immuno depression or immunodeficiency acquired or congenital
* Immuno depressor or corticoid treatments

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Number of infectious episodes | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc Cazaubiel, Dr, Principal Investigator — BioFortis
Locations (1):
- Biofortis, Nantes, France